CLINICAL TRIAL: NCT03564548
Title: Inhaled PPP001 Versus Immediate-release Oral Opioids for the Management of Breakthrough Pain in Cancer Subjects: a Randomized, Open Label, Crossover, Comparison Study
Brief Title: Inhaled Cannabinoids Versus Immediate-release Oral Opioids for the Management of Breakthrough Cancer Pain
Acronym: REBORN
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tetra Bio-Pharma (Industry)
Collaborators: Cognitive Research Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: PPP001-Ph2-03
Record Dates: First submitted 2018-05-22; First posted 2018-06-21 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Cancer; Breakthrough Cancer Pain
MeSH Terms: conditions — Neoplasms | interventions — Morphine; Hydromorphone; Oxycodone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PPP001 (Experimental): Inhaled cannabinoids (PPP001)
  Interventions: Drug: PPP001
- Morphine sulfate or Hydromorphone or Oxycodone (Active Comparator): Oral morphine sulfate or hydromorphone or oxycodone at the previous stabilized dosage
  Interventions: Drug: Morphine sulfate or Hydromorphone or Oxycodone

INTERVENTIONS:
Drug: PPP001 — Group assigned to PPP001
  Arms: PPP001
Drug: Morphine sulfate or Hydromorphone or Oxycodone — Group assigned to morphine sulfate or hydromorphone or oxycodone
  Arms: Morphine sulfate or Hydromorphone or Oxycodone

SUMMARY:
Breakthrough cancer pain (BTcP) is a rapid onset, high intensity and short duration pain episode, which takes place within stable background pain control. It significantly affects the quality of life of patients with cancer and their ability to function normally. Rapid onset opioids and immediate-release oral opioids (e.g. morphine sulfate, hydromorphone, and oxycodone) are the standard treatment for BTcP. Because of the limited availability, high cost, complicated titration and the high risks of overdosing with rapid-onset opioids, most often the preferred choice of treatment is immediate-release oral opioids. However, this approach might not always offer optimal speed for onset of action and duration to match the rapid nature of an episode of BTcP. In order to seek a potential alternative to immediate-release oral opioids, we are proposing to test the onset of action of PPP001 to rapidly alleviate breakthrough pain in patients with cancer. We will also examine the safety and the efficacy on pain intensity of PPP001 within this population.

DETAILED DESCRIPTION:
The study is a randomized, open-label crossover comparison study: This will be a 10-week open-label randomized study to evaluate the effect of inhaled PPP001 as compared to morphine sulfate or hydromorphone or oxycodone to improve for the treatment of BTcP. After proper screening and verified inclusion/exclusion criteria, 20 consecutive subjects will be recruited.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent.
2. Adult male and female subjects at least 18 years of age.
3. Subject agrees to follow the protocol.
4. Confirmed diagnosis of cancer with life expectancy of more than 3 months; Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2.
5. If currently receiving chemotherapy and/or radiotherapy treatment, subjects must be on a stable regimen for at least one month (30 days ± 2 days) prior to screening.
6. Background cancer pain stable (pain <4/10 on numeric rating scale) and adequately controlled with long-acting oral morphine, oxycodone, hydromorphone, hydrocodone, or meperidine.
7. Subject receiving at least 30 mg of oral morphine equivalent daily doses (MEDD) for both background and breakthrough cancer pain.
8. The subject is currently taking chronic treatment with opiod analgesic but still has a clinical diagnosis of breakthrough cancer pain with <3 episodes per day but >3 episodes per week.
9. The subject is using only oral morphine sulfate for breakthrough opioid analgesia.
10. Normal cognitive status according to MiniCog.
11. The subject is able to perform deep inhalations with FEV1 more than 60%.
12. Ability to read and respond to questions in English.
13. A female subject must meet one of the following criteria:

    If of childbearing potential - agrees to use one of the accepted contraceptive regimens from at least 28 days prior to the first drug administration, during the study and for at least 60 days after the last dose.

    If of non-childbearing potential - should be surgically sterile or in a menopausal state
14. A male subject with sexual partners who are pregnant, possibly pregnant, or who could become pregnant must be surgically sterile or agrees to use one of the accepted contraceptive regimens from first drug administration until 3 months after the last drug administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-05-26 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Time weighted Sum of Pain Intensity Differences from 0 to 30 minutes (SPID30). | change between 0 min (before starting treatment) and 30 minutes after dosing
  SPID30 score after PPP001 administration or immediate-release oral opioids (morphine sulfate or hydromorphone or oxycodone) administration. The SPID30 calculation is based on a 100 mm pain intensity VAS were 0 mm is the minimum and 100 mm the maximum with higher score representing a worse outcome.

SECONDARY OUTCOMES:
SPID at 10, 15, and 60 minutes | 10, 15, and 60 minutes after dosing
  SPID score after PPP001 administration or immediate-release oral opioids (morphine sulfate or hydromorphone or oxycodone) administration. The SPID calculation is based on a 100 mm pain intensity VAS were 0 mm is the minimum and 100 mm the maximum with higher score representing a worse outcome.
Pain intensity difference (PID) | 5, 10, 15, 30 and 60 minutes after dosing
  PID score after PPP001 administration or immediate-release oral opioids (morphine sulfate or hydromorphone or oxycodone) administration. The PID calculation is based on a 100 mm pain intensity VAS were 0 mm is the minimum and 100 mm the maximum with higher score representing a worse outcome.
Pain relief at 5, 10, 15, 30 and 60 minutes | 5, 10, 15, 30 and 60 minutes after dosing
  Subjective pain relief evaluated with a self-administered scale. The pain relief is measured with a five-point scale (0 = none to 4 = complete relief) with a higher score representing a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Hassman, Principal Investigator — Hassman Research Institute
Locations (1):
- HRI, Berlin, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided